CLINICAL TRIAL: NCT07032025
Title: A Prospective, Multicenter, Randomized Controlled Trial of the Catheter-directed Mechanical Thrombectomy Compared to Standard Anticoagulation for Use in the Treatment of Acute Intermediate-risk Pulmonary Embolism.
Brief Title: Mechanical Thrombectomy for Acute Pulmonary Embolism
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jun Pu, Professor, Chief Physician, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EARLY-MYO-PE
Record Dates: First submitted 2025-06-13; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Acute Pulmonary Embolism
Keywords: Prospective Studies; Pulmonary Embolism; Thrombectomy
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Innovative Device Group: Minimally invasive thrombectomy (Experimental)
  Interventions: Procedure: Innovative Device Group
- Standard Pharmacological Therapy Group: Pharmacological thrombolysis + anticoagulation (Active Comparator)
  Interventions: Drug: Standard Pharmacological Therapy Group

INTERVENTIONS:
Procedure: Innovative Device Group — Catheter-based thrombectomy is performed within 4 hours after baseline CTPA acquisition. Pre-procedural anticoagulation with either low-molecular-weight heparin (LMWH) or unfractionated heparin (UFH) is administered prior to thrombectomy. Post-procedural oral anticoagulation is transitioned to rivaroxaban 20 mg once daily (QD).
  Arms: Innovative Device Group: Minimally invasive thrombectomy
Drug: Standard Pharmacological Therapy Group — Following thrombolytic agent administration, anticoagulation with rivaroxaban is initiated and maintained at 15 mg twice daily (BID) for the initial 3 weeks, then switched to 20 mg once daily (QD) thereafter.
  Arms: Standard Pharmacological Therapy Group: Pharmacological thrombolysis + anticoagulation

SUMMARY:
Research Objective:

To prospectively compare the efficacy and safety of a pre-collaboratively developed ultra-thin PTFE minimally invasive thrombectomy system versus standard pharmacological therapy in patients with acute pulmonary embolism (PE), both administered on top of standard care.

Research Content:

Patients meeting all the following criteria will be enrolled:

Aged 18-75 years (male or female)

Clinically diagnosed with acute PE

Right ventricular/left ventricular diameter ratio (RV/LV) ≥0.9 on computed tomographic pulmonary angiography (CTPA)

Provision of voluntary written informed consent.

Study Design:

After confirming eligibility, subjects will be randomized at a 1:1 ratio into two groups:

Innovative Device Group: Minimally invasive thrombectomy

Standard Pharmacological Therapy Group: Pharmacological thrombolysis + anticoagulation

Study Endpoints:

Primary Efficacy Endpoint:

Reduction in RV/LV ratio (measured by CTPA) from baseline to 48 hours post-treatment.

Primary Safety Endpoint:

Incidence of Major Adverse Events (MAEs) from baseline to 48 hours post-treatment, defined as:

Procedure-related death

Major bleeding (per VARC-2 criteria: life-threatening, disabling, or major bleeding)

Treatment-related clinical deterioration, including:

Unplanned mechanical ventilation

Arterial hypotension (systolic blood pressure <90 mmHg for >1 hour or requiring vasopressors) or shock

Cardiopulmonary resuscitation

Sustained deterioration in oxygenation

Emergency surgical embolectomy.

Key Terminology Notes:

RV/LV: Right Ventricular/Left Ventricular diameter ratio (standard medical abbreviation retained).

VARC-2: Valve Academic Research Consortium-2 (internationally recognized bleeding criteria).

PTFE: Polytetrafluoroethylene (material name preserved).

MAE: Major Adverse Events (acronym defined at first use).

Clinical deterioration: Explicitly specified with objective clinical indicators.

This translation maintains scientific precision while adhering to international clinical trial reporting standards (ICH-GCP). The structure aligns with typical English-language study protocols for clarity and reproducibility.

DETAILED DESCRIPTION:
1. Research Objective To prospectively evaluate the comparative efficacy and safety of a novel ultra-thin polytetrafluoroethylene (PTFE) minimally invasive thrombectomy system versus guideline-directed pharmacological thrombolysis in patients with acute intermediate-high-risk pulmonary embolism (PE), both administered as adjuncts to standard anticoagulation therapy.
2. Study Population

   Inclusion Criteria:

   Adults aged 18-75 years (all genders)

   Acute PE confirmed by computed tomographic pulmonary angiography (CTPA) within 14 days of symptom onset

   Right ventricular dysfunction defined as RV/LV diameter ratio ≥0.9 on baseline CTPA

   Provision of written informed consent

   Exclusion Criteria:

   Absolute contraindications to thrombolysis (e.g., active bleeding, recent intracranial hemorrhage, major surgery within 14 days)

   Hemodynamic instability requiring immediate rescue therapy (systolic BP <90 mmHg with end-organ hypoperfusion)

   Severe renal impairment (eGFR <30 mL/min/1.73m²) or hepatic failure (Child-Pugh Class C)

   Life expectancy <6 months due to non-PE comorbidities
3. Study Design Design: Prospective, multicenter, open-label, randomized controlled trial with blinded endpoint adjudication

   Randomization: Eligible subjects stratified by PE severity (RV/LV: 0.9-1.0 vs. >1.0) and thrombus burden (main/lobar vs. segmental PA involvement), then randomized 1:1 via centralized web-based system.

   Intervention Groups:

   Group A (Innovative Device):

   Ultra-thin PTFE thrombectomy catheter deployed under fluoroscopic guidance via femoral access

   Procedure completion within 90 minutes; mandatory peri-procedural unfractionated heparin (target ACT 250-300 s)

   Post-procedure: Enoxaparin 1 mg/kg BID → transitioned to rivaroxaban 20 mg OD at 24 hours

   Group B (Standard Therapy):

   Alteplase infusion: 10 mg bolus + 90 mg over 2 hours (max 100 mg)

   Concurrent heparin infusion (target aPTT 60-80 s) → switched to rivaroxaban 15 mg BID (Day 1-21) → 20 mg OD thereafter
4. Endpoint Definitions Primary Efficacy Endpoint Absolute reduction in RV/LV ratio from baseline to 48 hours post-intervention, measured by blinded core-lab CTPA analysis.

   Primary Safety Endpoint

   Composite Major Adverse Events (MAEs) within 48 hours, including:

   Procedure-related mortality

   Major bleeding per VARC-2 criteria:

   Fatal bleeding

   Intracranial hemorrhage

   Bleeding causing ≥3 g/dL hemoglobin drop or transfusion of ≥2 units

   Bleeding requiring surgical intervention

   Treatment-related clinical deterioration:

   Unplanned mechanical ventilation

   Sustained hypotension (SBP <90 mmHg for >1 hour requiring vasopressors)

   Cardiopulmonary resuscitation

   New requirement for ECMO or emergency surgical embolectomy
5. Statistical Analysis Plan

   Sample Size: 142 subjects/group (total N=284) providing 90% power (α=0.05) to detect:

   Efficacy: Mean RV/LR reduction difference of 0.15 (SD=0.3)

   Safety: 40% relative risk reduction in MAEs (Group A: 10% vs. Group B: 17%)

   Analysis Sets:

   Primary analysis: Modified intention-to-treat (mITT; all randomized receiving ≥1 treatment component)

   Safety analysis: As-treated population

   Methods:

   Continuous variables: Mixed-effects repeated measures ANOVA

   Categorical variables: Cochran-Mantel-Haenszel test with stratification adjustment

   Time-to-event: Kaplan-Meier with log-rank test
6. Quality Assurance Endpoint Adjudication Committee: Blinded to treatment allocation

Data Monitoring: Independent DSMB reviewing unblinded safety data quarterly

Procedure Standardization:

All interventionalists certified via simulation training (≥5 proctored cases)

Centralized core lab for CTPA RV/LV measurements

Ethical Compliance: Approved by institutional review boards at all sites (NCT# pending). Trial conducted per Declaration of Helsinki.

Key Advantages of Expanded Protocol Stratified randomization controls confounding from baseline RV strain heterogeneity.

VARC-2 bleeding criteria enhance comparability with cardiovascular intervention trials.

Core-lab blinded CTPA analysis eliminates measurement bias in efficacy assessment.

Pre-specified safety triggers (e.g., Hb drop thresholds) enable objective MAE classification.

Standardized anticoagulation bridging minimizes post-procedural thrombotic risk variability.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years (male or female)
* Clinically diagnosed with acute PE
* Right ventricular/left ventricular diameter ratio (RV/LV) ≥0.9 on computed tomographic pulmonary angiography (CTPA)
* Provision of voluntary written informed consent.

Exclusion Criteria:

* Target vessel diameter <6 mm
* Calcification, plaque, or stenosis in target lesion
* Sustained systolic blood pressure <90 mmHg for >15 minutes or requiring vasopressors to maintain SBP ≥90 mmHg
* Peak pulmonary artery pressure >70 mmHg
* Hematocrit <28%
* History of chronic pulmonary hypertension
* Pre-existing left bundle branch block
* Chronic left heart failure with left ventricular ejection fraction (LVEF) ≤30%
* Renal dysfunction (serum creatinine >1.8 mg/dL or >159 μmol/L)
* Known coagulopathy or bleeding diathesis:

Platelet count <50×10⁹/L, or International Normalized Ratio (INR) >3

* Contraindications to antiplatelet/anticoagulant therapy
* Cardiothoracic or pulmonary surgery within 7 days prior
* Intracardiac thrombus
* Patients on extracorporeal membrane oxygenation (ECMO)
* Known hypersensitivity to iodinated contrast media
* Significant comorbidities complicating treatment/evaluation:

Active malignancy Acute infectious disease/sepsis Systemic conditions precluding procedure tolerance Life expectancy <1 year

* Pregnant or lactating women
* Concurrent participation in other drug/device trials
* Other investigator-determined unsuitability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | 48 hours post-treatment.
  Reduction in RV/LV ratio (measured by CTPA) from baseline to 48 hours post-treatment.
Primary Safety Endpoint: | 48 hours post-treatment
  Incidence of Major Adverse Events (MAEs) from baseline to 48 hours post-treatment